CLINICAL TRIAL: NCT02153632
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind, 26 Week Study to Evaluate the Efficacy and Safety of Amantadine HCl Extended Release Tablets in Parkinson's Disease Subjects With Levodopa-Induced Dyskinesias
Brief Title: Efficacy and Safety of Amantadine Hydrogen Chloride (HCl) ER Tablets in Parkinson's Disease Subjects With LID
Acronym: ALLAY-LID-II
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Adamas Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OS320-3006
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Parkinson's Disease; Levodopa Induced Dyskinesia (LID)
Keywords: Parkinson's Disease; Levodopa Induced Dyskinesia (LID); LID; Parkinsonism; Dyskinesia
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Dyskinesias | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 240mg amantadine HCl ER tablets (Experimental): amantadine HCl ER, 240 mg tablets, once daily, 22 weeks
  Interventions: Drug: amantadine HCl ER
- 320mg amantadine HCl ER tablets (Experimental): amantadine HCl ER, 320 mg tablets, once daily, 22 weeks
  Interventions: Drug: amantadine HCl ER
- Placebo Tablets for Amantadine (Placebo Comparator): Placebo, tablets, once daily, 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: amantadine HCl ER — Subjects are given either 240 mg amantadine HCl ER tablet or 320 mg amantadine HCl ER tablet
  Other Names: Osmolex ER Tablet
  Arms: 240mg amantadine HCl ER tablets; 320mg amantadine HCl ER tablets
Drug: Placebo — subjects are given an identical placebo tablet
  Other Names: Placebo tablets
  Arms: Placebo Tablets for Amantadine

SUMMARY:
The purpose of this multi-center, randomized, double-blind, parallel-group, 26 week study is to compare the efficacy and safety of two different dose levels of Amantadine Extended Release Tablets to placebo for the treatment of levodopa induced dyskinesia in patients with Parkinson's disease.

DETAILED DESCRIPTION:
This study was terminated early due to slow enrollment with 135 of 162 planned subjects enrolled. Amantadine HCl ER has been used for many years as a treatment for Parkinson's disease. It has been reported in the literature to effectively treat the motor complications of levodopa, especially dyskinesia, but it must be given 2 to 4 times a day. The purpose of this multi-center, randomized, double-blind, parallel-group, 26 week study is to compare the efficacy and safety of two different dose levels of Amantadine Extended Release Tablets to placebo for the treatment of levodopa induced dyskinesia in patients with Parkinson's disease. The dose will be given once a day in the morning so that amantadine concentrations are maintained throughout the day for treating the levodopa induced dyskinesia, but will be lower during the night, potentially reducing the negative impact of amantadine on sleep.

ELIGIBILITY:
Inclusion Criteria:

* Signed Institutional Review Board (IRB)/ Independent Ethics Committee (IEC) informed consent form.
* Idiopathic Parkinson's disease per the United Kingdom (UK) Parkinson's Disease Society Brain Bank criteria.
* Male or female 30 to 85 years old.
* Levodopa induced, predictable peak-effect dyskinesia considered problematic and/or disabling.
* Screening serum creatinine level within normal range
* On stable doses of all oral anti-Parkinson's medication, including any levodopa preparation, for 30 days and be willing to remain on the same doses throughout the trial.
* The subject/caregiver must demonstrate the ability to complete an accurate home diary based on training and evaluation during the screening period.

Exclusion Criteria:

* Secondary parkinsonian syndrome, such as vascular, postinflammatory,drug-induced, neoplastic and post-traumatic parkinsonism or any atypical parkinsonian syndrome (e.g., Progressive Supranuclear Palsy, Multi-System Atrophy, etc.);
* Use of amantadine within 14 days before study start, or previously had an adverse event to amantadine
* Currently taking neuroleptics and atypical antipsychotic agents, acetylcholinesterase inhibitors, apomorphine, rimantadine, memantine and dextromethorphan and quinidine if used in combination for treating dyskinesia.
* History of neurosurgical intervention for treating Parkinson's s disease (i.e. pallidotomy or implanted with a deep brain stimulator)
* Any medical condition or past medical history that would increase the risk of exposure to Amantadine HCl Extended Release Tablets or interfere with safety and efficacy evaluations.
* History of cancer within 5 years of screening with following exceptions: adequately treated non-melanomatous skin cancers, localized bladder cancer, non-metastatic prostate cancer or in situ cervical cancer.
* History or current diagnosis of schizophrenia or bipolar disorder;
* Inadequately treated Major Depressive Disorder. Subjects on stable doses of selective serotonin reuptake inhibitors (SSRIs) or serotonin-norepinephrine reuptake inhibitors (SNRIs) are eligible for the study;
* Is at imminent risk of suicide or had a suicide attempt within 6 months of screening
* History or current diagnosis of Impulse Control Disorder
* Calculated plasma creatinine clearance of <60 mL/min at screening
* History of or currently has any of the following clinically significant conditions, cardiovascular, respiratory, renal, hepatic, or gastrointestinal disease
* Any clinically significant vital sign, ECG, or laboratory abnormalities;
* A positive test for HIV antibody or history of HIV; hepatitis B surface antigen unless the positive test followed a recent (<28 days) vaccination for hepatitis B; hepatitis C antibody;
* A positive urine drug test.
* Pregnant or breastfeeding at screening or has a positive pregnancy test
* If a sexually active female, is not surgically sterile or at least 2 years post-menopausal, or does not agree to utilize an effective method of contraception from the screening visit to at least 4 weeks after the completion of study treatment.
* History of alcohol or narcotic substance abuse ≤1 year before screening.
* Has dementia or another psychiatric illness that prevents provision of informed consent.
* Has a known hypersensitivity to the study treatment(s), based on known allergies to drugs of the same class including rimantadine HCl and memantine HCl.
* Has participated in other studies involving investigational drugs or surgeries within the last 30 days or investigational biologics within the last 6 months prior to screening.
* Plans to undergo major elective surgery during the course of the study.
* Received administration of Live Attenuated Influenza Vaccine (LAIV) within 2 weeks.
* Cognitive impairment, as evidenced by a score <26 on the Montreal Cognitive Assessment (MoCA) at the screening visit.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dentiste, MBA, Study Chair — Osmotica Pharmaceutical US LLC
Locations (56):
- United States (24):
  - Tucson, Arizona
  - Fountain Valley, California
  - Irvine, California
  - Pasadena, California
  - Ventura, California
  - Boulder, Colorado
  - Hollywood, Florida
  - Miami, Florida
  - North Palm Beach, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Ann Arbor, Michigan
  - Summit, New Jersey
  - Brooklyn, New York
  - Patchogue, New York
  - Raleigh, North Carolina
  - Columbus, Ohio
  - Round Rock, Texas
  - Orem, Utah
  - Kirkland, Washington
- Ottawa, Ontario, Canada
- France (12):
  - Rennes, Ille Et Vilaine
  - Amiens
  - Bron
  - Clermont-Ferrand
  - Créteil
  - Lille
  - Marseille
  - Montauban
  - Nîmes
  - Paris
  - Poitiers
  - Toulouse
- Germany (9):
  - Haag, Bavaria
  - Erbach im Odenwald, Hesse
  - Achim, Niedersachesen
  - Bochum, North Rhine-Westphalia
  - Hindenburg, State of Berlin
  - Weissensee, State of Berlin
  - Berlin
  - Wiesbaden
  - Würzburg
- Spain (10):
  - L'Hospitalet de Llobregat, Barcelona
  - Manresa, Barcelona
  - Seville, Barcelona
  - Vallés, Barcelona
  - Alcorcón, Madrid
  - Castellana, Madrid
  - Marañón, Madrid
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General de Cataluna, Barcelona
  - Pamplona

RESULTS

PARTICIPANT FLOW:
Groups:
- 240mg Amantadine HCl ER Tablets: Amantadine Hydrogen Chloride (HCl) ER Tablets 240mg daily for 22 weeks post two week titration phase.
  Amantadine HCl ER (ALLAY-LID II)
- 320mg Amantadine HCl ER Tablets: Amantadine HCl ER Tablets 320mg daily for 22 weeks post two week titration phase.
  Amantadine HCl ER (ALLAY-LID II)
- Placebo Tablets for Amantadine: Placebo Tablets matching Amantadine HCl ER Tablets taken daily for 26 weeks.
  Placebo
Period: Overall Study
Arm/Group | 240mg Amantadine HCl ER Tablets | 320mg Amantadine HCl ER Tablets | Placebo Tablets for Amantadine
Started | 45 | 46 | 44
Completed | 27 | 27 | 25
Not Completed | 18 | 19 | 19

BASELINE CHARACTERISTICS:
Groups:
- 240mg Amantadine HCl ER Tablets: Amantadine HCl ER Tablets 240mg daily for 22 weeks post two week titration phase.
  Amantadine HCl ER (ALLAY-LID II)
- Total: Total of all reporting groups
Arm/Group | 240mg Amantadine HCl ER Tablets | 320mg Amantadine HCl ER Tablets | Placebo Tablets for Amantadine | Total
Number analyzed (Participants) | 45 | 46 | 44 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 46 | 44 | 135
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.88) | 63.0 (8.98) | 63.5 (10.36) | 63.5 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 18 | 55
  Male | 29 | 25 | 26 | 80
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 1 | 2 | 6
  United States | 15 | 23 | 23 | 61
  France | 10 | 7 | 8 | 25
  Germany | 7 | 6 | 6 | 19
  Spain | 10 | 9 | 5 | 24

OUTCOME MEASURES:

1. Primary Outcome: Unified Dyskinesia Rating Scale
Description: The Unified Dyskinesia Rating Scale is a validated tool for assessment of dyskinesia (involuntary movements) in Parkinson's Disease patients. Rating consists of the change from baseline to Day 98 of the sum of the 26 questions comprising the questionnaire. Each question in the questionnaire is rated on a 5 point scale from 0-4 where 0 is a better outcome. Questions assess: over the past week total hours with dyskinesia and total hours without dyskinesia; problems with speech, chewing and swallowing, eating, dressing, hygiene, handwriting, hobbies, balance, socializing, emotions, spasm or cramps, pain without dystonia and pain from dystonia. The minimum (better) value is 0 and the maximum (worse) value is 130.
Time Frame: Change from baseline to Day 98
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 240mg Amantadine HCl ER Tablets | 320mg Amantadine HCl ER Tablets | Placebo Tablets for Amantadine
Number analyzed (Participants) | 45 | 46 | 44
score on a scale
  Visit 2 (Baseline): number analyzed (Participants) | 44 | 45 | 44
  Visit 2 (Baseline) | 41.3 (13.91) | 36.3 (12.40) | 40.7 (13.98)
  Visit 7 (Day 98)/Stable Dose LOCF [1]: number analyzed (Participants) | 41 | 43 | 37
  Visit 7 (Day 98)/Stable Dose LOCF [1] | 41.3 (13.98) | 36.3 (12.40) | 40.7 (13.98)
  Mean Change from Baseline (SD): number analyzed (Participants) | 41 | 43 | 37
  Mean Change from Baseline (SD) | -15.2 (15.58) | -13.7 (10.95) | -9.0 (10.62)
Statistical Analysis 1: Comparison: 240mg Amantadine HCl ER Tablets; Test type: Superiority; p = 0.031, ANCOVA; Mean Difference (Final Values) = -5.5, 95% CI 2-sided [-10.5 to -0.5], Standard Error of Mean 1.75
Statistical Analysis 2: Comparison: 320mg Amantadine HCl ER Tablets; Test type: Superiority; p = 0.011, ANCOVA; Mean Difference (Final Values) = -6.5, 95% CI 2-sided [-11.5 to -1.5], Standard Error of Mean 1.71

2. Secondary Outcome: Mobility State Self-Assessment - Subject Diary Cards
Description: hange from baseline in the number of awake hours without troublesome dyskinesia (involuntary movements). Every half hour the subject will indicate in the diary if the medication has ("ON") or has not ("OFF") produced benefits in terms of mobility, slowness and rigidity. Valid diaries of the 3 consecutive days prior to each visit will be averaged with respect to the number of awake hours without troublesome dyskinesia. The change from baseline in the number of waking hours that subjects report being "ON" without troublesome dyskinesias will be analyzed at analysis visits Day 14 and Day 98 of treatment. Higher scores mean a better outcome and the maximum value is 24 hours.
Time Frame: Day 14 and Day 98 of treatment
Population: The number analyzed is the number of subjects with values at each time point.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 240mg Amantadine HCl ER Tablets | 320mg Amantadine HCl ER Tablets | Placebo Tablets for Amantadine
Number analyzed (Participants) | 45 | 46 | 44
Hours
  Visit 2 (Baseline): number analyzed (Participants) | 43 | 45 | 39
  Visit 2 (Baseline) | 10.4 (3.76) | 9.8 (3.48) | 9.1 (3.48)
  Visit 7 (Day 98)/Stable Dose LOCF [1] | 12.7 (3.91) | 13.3 (3.83) | 11.1 (4.03)
  Mean Change in Hours from Baseline (SD) | 2.3 (3.25) | 3.6 (3.93) | 1.6 (3.56)

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | 240mg Amantadine HCl ER Tablets | 320mg Amantadine HCl ER Tablets | Placebo Tablets for Amantadine
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/46 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/45 | 4/46 | 6/44
Other Adverse Events (participants affected / at risk) | 36/45 | 38/46 | 29/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 240mg Amantadine HCl ER Tablets (N=45) | 320mg Amantadine HCl ER Tablets (N=46) | Placebo Tablets for Amantadine (N=44)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
constipation hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
cranial nerve palsies multiple (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
contipation diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 240mg Amantadine HCl ER Tablets (N=45) | 320mg Amantadine HCl ER Tablets (N=46) | Placebo Tablets for Amantadine (N=44)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 5 (5) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 4 (4)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod sting (General disorders) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 5 (5) | 3 (3)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | 5 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Chloesterol increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine renal clearance increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Crystal urine present (Investigations) | 1 (1) | 2 (2) | 1 (1)
Electrocardiogram QT Shortened (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocadiogram T wave abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin urine present (Investigations) | 1 (1) | 3 (3) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Mean cell hemoglobin concentration decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Red blood cells urine positive (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary casts present (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urine ketone body present (Investigations) | 1 (1) | 1 (1) | 0 (0)
Urine leukocyte esterase positive (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 2 (2) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Food Craving (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
muscle spasm (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1)
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Temporomandibular join syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Action tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Akinesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Bradykinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Circadian rhythm sleep disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cranial nerve palsies multiple (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 5 (5) | 3 (3) | 3 (3)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Freezing phenomenon (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Mental impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Parkinson's disease (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 3 (3) | 0 (0) | 4 (4)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Hallucination (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 3 (3) | 2 (2) | 1 (1)
Hallucinations, mixed (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Illusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Impulsive behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Libido increased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Middle insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Rapid eye movements sleep abnormal (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Sleep attacks (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1) | 2 (2)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Varicophebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall allow SPONSOR 60 days to review any manuscript and 30 days to review any poster presentation, abstract or any other written or oral material which discloses the Study Results. SPONSOR may request in writing an additional 60 days for review.

SPONSOR may remove all Confidential Information from any publications or presentations, or if deemed not sufficient to protect its Intellectual Property Rights, then SPONSOR may embargo the publication or presentation.